CLINICAL TRIAL: NCT00846365
Title: A Phase 3, Double-Blind, Randomized, Efficacy and Safety Study Comparing the TAK-491 Plus Chlorthalidone Fixed-Dose Combination vs Benicar HCT® (Olmesartan Medoxomil-Hydrochlorothiazide) in Subjects With Moderate to Severe Essential Hypertension
Brief Title: Efficacy and Safety of Azilsartan Medoxomil Plus Chlorthalidone in Participants With Moderate to Severe Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAK-491CLD_301; U1111-1112-4287 (Other: WHO)
Record Dates: First submitted 2009-02-13; First posted 2009-02-18 (Estimated); Results first posted 2012-03-13 (Estimated); Last update posted 2012-03-13 (Estimated); Status verified 2012-02

CONDITIONS: Essential Hypertension
Keywords: Essential Hypertension; Hypertensive; Blood Pressure, High; Vascular Disease; Cardiovascular Disease; Drug Therapy
MeSH Terms: conditions — Essential Hypertension; Hypertension; Vascular Diseases; Cardiovascular Diseases | interventions — azilsartan medoxomil; Chlorthalidone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Azilsartan Medoxomil 20-40mg plus Chlorthalidone 12.5-25 mg QD (Experimental): (dependant on blood pressure)
  Interventions: Drug: Azilsartan medoxomil and chlorthalidone
- Azilsartan Medoxomil 40-80mg plus Chlorthalidone 12.5-25 mg QD (Experimental): (dependant on blood pressure)
  Interventions: Drug: Azilsartan medoxomil and chlorthalidone
- Olmesartan medoxomil 20-40mg/hydrochlorothiazide 12.5-25mg QD (Active Comparator): (dependant on blood pressure)
  Interventions: Drug: Olmesartan medoxomil-hydrochlorothiazide

INTERVENTIONS:
Drug: Azilsartan medoxomil and chlorthalidone — Azilsartan medoxomil 20 mg and chlorthalidone 12.5 mg, tablets, orally, and olmesartan medoxomil-hydrochlorothiazide placebo tablets once daily for 8 weeks.
  If participant does not achieve target blood pressure at Week 4, then the dosage will be increased to azilsartan medoxomil 40 mg and chlorthalidone 25 mg, tablets, orally, once daily for the remaining 4 weeks.
  Other Names: azilsartan medoxomil; chlorthalidone; TAK-491; TAK-491CLD
  Arms: Azilsartan Medoxomil 20-40mg plus Chlorthalidone 12.5-25 mg QD
Drug: Azilsartan medoxomil and chlorthalidone — Azilsartan medoxomil 40 mg and chlorthalidone 12.5, mg, tablets, orally, and olmesartan medoxomil-hydrochlorothiazide placebo tablets once daily for 8 weeks.
  If participant does not achieve target blood pressure at Week 4, then the dosage will be increased to azilsartan medoxomil 80 mg and chlorthalidone 25 mg, tablets, orally, once daily for the remaining 4 weeks.
  Other Names: azilsartan medoxomil; chlorthalidone; TAK-491; TAK-491CLD
  Arms: Azilsartan Medoxomil 40-80mg plus Chlorthalidone 12.5-25 mg QD
Drug: Olmesartan medoxomil-hydrochlorothiazide — Olmesartan medoxomil 20 mg/hydrochlorothiazide 12.5 mg, tablets, orally, and Azilsartan medoxomil and chlorthalidone placebo-matching tablets, orally, once daily for 8 weeks.
  If participant does not achieve target blood pressure at Week 4, then the dosage will be increased to olmesartan medoxomil 40 mg/hydrochlorothiazide 25 mg, tablets, orally, once daily for the remaining 4 weeks.
  Other Names: Benicar HCT®
  Arms: Olmesartan medoxomil 20-40mg/hydrochlorothiazide 12.5-25mg QD

SUMMARY:
The purpose of this study is to determine the efficacy and safety of azilsartan medoxomil combined with chlorthalidone, once daily (QD), in participants with moderate to severe essential hypertension.

DETAILED DESCRIPTION:
According to the World Health Organization, hypertension is the most common attributable cause of preventable death in developed nations, as uncontrolled hypertension greatly increases the risk of cardiovascular disease, cerebrovascular disease and renal failure. As the population ages, the prevalence of hypertension will continue to increase if broad and effective preventive measures are not implemented. Despite the availability of antihypertensive agents, hypertension remains inadequately controlled; only about one-third of patients continue to maintain control successfully.

Although most antihypertensive agents are effective at the appropriate dose, the majority have side effects that limit their use. As a class, angiotensin II receptor blockers generally are considered more tolerable than other classes of antihypertensive agents. TAK-491 (azilsartan medoxomil) is an angiotensin II receptor blocker being evaluated by Takeda to treat essential hypertension.

Treatments for essential hypertension commonly include use of a thiazide-like diuretic, either alone or as part of combination treatment. Although chlorthalidone was commonly prescribed in the past, its use has widely been replaced with hydrochlorothiazide, presumably due to a lack of available combination products containing chlorthalidone, the assumption that hydrochlorothiazide and chlorthalidone have similar antihypertensive effects and cardiovascular benefits, and the perception that chlorthalidone use is associated with a greater frequency of hypokalemia. However, the frequency of hypokalemia with chlorthalidone use is relatively low in the dose range of 12.5 to 25 mg and these doses have been shown to be associated with potent blood pressure reduction. Several long-term outcomes trials have shown that blood pressure reductions associated with chlorthalidone treatment reduce risk of cardiovascular morbidity and mortality.

Most hypertensive patients require two or more agents to achieve target blood pressure and diuretics are commonly used in combination with other antihypertensive agents.

Participants in this study will be randomized to receive one of 3 possible dosing combinations of azilsartan medoxomil with either chlorthalidone or olmesartan medoxomil-hydrochlorothiazide over 8 weeks. The total duration of the study is approximately 13 weeks. Participants will make a total of 11 visits to the clinic, and will be required to participate in a follow-up telephone call 14 days after last dose of the study drug for adverse event assessment.

ELIGIBILITY:
Inclusion Criteria:

1. 190 mm Hg on Day -1 or if the participant has not received antihypertensive treatment within 28 days before screening and has a mean sitting clinic systolic blood pressure greater than or equal to 160 and less than or equal to 190 mm Hg at the Screening Visit and on Day -1.
2. Females of childbearing potential who are sexually active must agree to use adequate contraception, and can neither be pregnant nor lactating from Screening throughout the duration of the study.
3. Has clinical laboratory test results within the reference range for the testing laboratory or the investigator does not consider the results to be clinically significant.
4. Is willing to discontinue current antihypertensive medications on Day -21 or on Day -28 if is on amlodipine or chlorthalidone.

Exclusion Criteria:

1. Has a mean sitting clinic diastolic blood pressure greater than 119 mm Hg.
2. Has a baseline 24-hour ambulatory blood pressure monitoring reading of insufficient quality.
3. Works a night (third) shift (from 11 PM [2300] to 7 AM [0700]).
4. Has an upper arm circumference less than 24 cm or greater than 42 cm.
5. Is noncompliant with study medication during the placebo run-in period.
6. Has secondary hypertension of any etiology.
7. Has a recent history of myocardial infarction, heart failure, unstable angina, coronary artery bypass graft, percutaneous coronary intervention, hypertensive encephalopathy, cerebrovascular accident or transient ischemic attack.
8. Has a clinically significant cardiac conduction.
9. Has hemodynamically significant left ventricular outflow obstruction due to aortic valvular disease.
10. Has severe renal dysfunction or disease.
11. Has a known or suspected unilateral or bilateral renal artery stenosis.
12. Has a history of cancer that has not been in remission for at least 5 years prior to the first dose of study drug.
13. Has poorly controlled type 1 or type 2 diabetes mellitus.
14. Has hypokalemia or hyperkalemia.
15. Has an alanine aminotransferase or aspartate aminotransferase level of greater than 2.5 times the upper limit of normal, active liver disease or jaundice.
16. Has any other known serious disease or condition that would compromise safety, might affect life expectancy or make it difficult to successfully manage and follow the participant according to the protocol.
17. Has a known hypersensitivity to angiotensin II receptor blockers or thiazide-type diuretics or other sulfonamide-derived compounds.
18. Has been randomized in a previous Azilsartan Medoxomil study.
19. Is currently participating in another investigational study or has participated in an investigational study or is receiving or has received any investigational compound within 30 days prior to Randomization.
20. Has a history of drug abuse or a history of alcohol abuse within the past 2 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1085 (Actual)
Dates: Start 2009-03; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Executive Medical Director, Study Director — Takeda
Locations (80):
- United States (70):
  - Birmingham, Alabama
  - Haleyville, Alabama
  - Hueytown, Alabama
  - Jasper, Alabama
  - Tallassee, Alabama
  - Green Valley, Arizona
  - Phoenix, Arizona
  - Long Beach, California
  - National City, California
  - Roseville, California
  - San Francisco, California
  - San Jose, California
  - Newark, Delaware
  - Clearwater, Florida
  - Jacksonville, Florida
  - Jupiter, Florida
  - Miami, Florida
  - Ocala, Florida
  - Pembroke Pines, Florida
  - Plant City, Florida
  - Tallahassee, Florida
  - Arlington Heights, Illinois
  - Chicago, Illinois
  - Gurnee, Illinois
  - Avon, Indiana
  - Wichita, Kansas
  - Louisville, Kentucky
  - Auburn, Maine
  - Baltimore, Maryland
  - Brockton, Massachusetts
  - Haverhill, Massachusetts
  - North Dartmouth, Massachusetts
  - Bingham Farms, Michigan
  - Stevensville, Michigan
  - Olive Branch, Mississippi
  - Kansas City, Missouri
  - New York, New York
  - Burlington, North Carolina
  - Charlotte, North Carolina
  - Hickory, North Carolina
  - Shelby, North Carolina
  - Akron, Ohio
  - Cleveland, Ohio
  - Columbus, Ohio
  - Marion, Ohio
  - Middleburg Heights, Ohio
  - Willoughby Hills, Ohio
  - Norman, Oklahoma
  - Bensalem, Pennsylvania
  - Erie, Pennsylvania
  - Reading, Pennsylvania
  - Cranston, Rhode Island
  - Cumberland, Rhode Island
  - North Charleston, South Carolina
  - Jackson, Tennessee
  - Kingsport, Tennessee
  - Milan, Tennessee
  - Austin, Texas
  - Corpus Christi, Texas
  - Dallas, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
  - Arlington, Virginia
  - Burke, Virginia
  - Charlottesville, Virginia
  - Manassas, Virginia
  - Lakewood, Washington
  - Port Orchard, Washington
  - Menomonee Falls, Wisconsin
- Chile (5):
  - Temuco, Cautín
  - La Serena, Elqui
  - Osorno, Osorno
  - Viña del Mar, Región de Valparaíso
  - Santiago, Santiago Metropolitan
- Mexico (5):
  - Chihuahua City, Chihuahua
  - Tijuana, Estado de Baja California
  - León, Guanajuato
  - Guadalajara, Jalisco
  - San Luis Potosí City, San Luis Potosí

REFERENCES:
- [Derived] Cushman WC, Bakris GL, White WB, Weber MA, Sica D, Roberts A, Lloyd E, Kupfer S. A randomized titrate-to-target study comparing fixed-dose combinations of azilsartan medoxomil and chlorthalidone with olmesartan and hydrochlorothiazide in stage-2 systolic hypertension. J Hypertens. 2018 Apr;36(4):947-956. doi: 10.1097/HJH.0000000000001647. PMID 29334491

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants enrolled at 93 investigative sites in Argentina, Chile, Mexico and the United States from 13 March 2009 to 25 June 2010.
Pre-assignment Details: Participants with moderate to severe essential hypertension were enrolled in one of 3, once-daily (QD) treatment groups.
Groups:
- Azilsartan Medoxomil 20-40mg Plus Chlorthalidone 12.5-25 mg QD: Azilsartan medoxomil 20 mg and chlorthalidone 12.5 mg, tablets, orally, and olmesartan medoxomil-hydrochlorothiazide placebo tablets once daily for 8 weeks.
  If participant does not achieve target blood pressure at Week 4, then the dosage will be increased to azilsartan medoxomil 40 mg and chlorthalidone 25 mg, tablets, orally, once daily for the remaining 4 weeks.
- Azilsartan Medoxomil 40-80mg Plus Chlorthalidone 12.5-25 mg QD: Azilsartan medoxomil 40 mg and chlorthalidone 12.5, mg, tablets, orally, and olmesartan medoxomil-hydrochlorothiazide placebo tablets once daily for 8 weeks.
  If participant does not achieve target blood pressure at Week 4, then the dosage will be increased to azilsartan medoxomil 80 mg and chlorthalidone 25 mg, tablets, orally, once daily for the remaining 4 weeks.
- Olmesartan Medoxomil 20-40mg/Hydrochlorothiazide 12.5-25mg QD: Olmesartan medoxomil 20 mg/hydrochlorothiazide 12.5 mg, tablets, orally, and Azilsartan medoxomil and chlorthalidone placebo-matching tablets, orally, once daily for 8 weeks.
  If participant does not achieve target blood pressure at Week 4, then the dosage will be increased to olmesartan medoxomil 40 mg/hydrochlorothiazide 25 mg, tablets, orally, once daily for the remaining 4 weeks.
Period: Overall Study
Arm/Group | Azilsartan Medoxomil 20-40mg Plus Chlorthalidone 12.5-25 mg QD | Azilsartan Medoxomil 40-80mg Plus Chlorthalidone 12.5-25 mg QD | Olmesartan Medoxomil 20-40mg/Hydrochlorothiazide 12.5-25mg QD
Started | 372 | 357 | 356
Completed | 317 | 308 | 323
Not Completed | 55 | 49 | 33
Not completed — Adverse Event | 20 | 30 | 11
Not completed — Protocol Violation | 5 | 4 | 0
Not completed — Lost to Follow-up | 8 | 2 | 5
Not completed — Withdrawal by Subject | 11 | 11 | 9
Not completed — Pregnancy | 1 | 0 | 0
Not completed — Lack of Efficacy | 1 | 1 | 2
Not completed — Other | 9 | 1 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Azilsartan Medoxomil 20-40mg Plus Chlorthalidone 12.5-25 mg QD | Azilsartan Medoxomil 40-80mg Plus Chlorthalidone 12.5-25 mg QD | Olmesartan Medoxomil 20-40mg/Hydrochlorothiazide 12.5-25mg QD | Total
Number analyzed (Participants) | 372 | 357 | 356 | 1085
Age Continuous [Mean (Standard Deviation); unit: years] | 55.5 (10.49) | 56.7 (10.83) | 55.7 (9.78) | 56.0 (10.38)
Age, Customized [Number; unit: participants]
  <45 years | 47 | 38 | 41 | 126
  45 to 64 years | 252 | 244 | 249 | 745
  ≥65 years | 73 | 75 | 66 | 214
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 175 | 174 | 173 | 522
  Male | 197 | 183 | 183 | 563
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Ethnicity was not collected from Latin American sites.
  Participants
    Hispanic or Latino | 37 | 41 | 44 | 122
    Not Hispanic or Latino | 265 | 253 | 251 | 769
    Unknown or Not Reported | 70 | 63 | 61 | 194
Race (NIH/OMB) [Number; unit: participants] — Participants could choose more than one category for race. Participants who chose more than 1 race category are included in each category indicated and are also included in the multiracial category.
  participants
    American Indian or Alaska Native | 37 | 34 | 35 | 106
    Asian | 7 | 5 | 5 | 17
    Native Hawaiian or Other Pacific Islander | 3 | 0 | 0 | 3
    Black or African American | 95 | 95 | 100 | 290
    White | 235 | 225 | 220 | 680
    More than one race | 5 | 2 | 4 | 11
    Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 302 | 294 | 295 | 891
  Mexico | 45 | 44 | 43 | 132
  Chile | 12 | 10 | 9 | 31
  Argentina | 13 | 9 | 9 | 31
Weight [Mean (Standard Deviation); unit: kg] | 89.35 (20.995) | 89.87 (21.281) | 90.66 (20.700) | 89.95 (20.981)
Height [Mean (Standard Deviation); unit: cm] | 167.5 (11.22) | 167.8 (11.06) | 168.2 (10.30) | 167.8 (10.87)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — BMI was calculated using height at Screening and weight at Baseline.
  kg/m^2 | 31.7 (5.94) | 31.8 (6.40) | 31.9 (6.08) | 31.8 (6.14)
Estimated Glomerular Filtration Rate (eGFR) Category [Number; unit: participants] — eGFR = creatinine clearance, estimated using the Modification of Diet in Renal Disease equation with the following parameters:
  * Moderate impairment: ≥30 to <60 mL/min/1.73 m^2
  * Mild impairment: ≥60 to <90 mL/min/1.73 m^2
  * Normal: ≥90 mL/min/1.73 m^2
  participants
    Moderate impairment | 26 | 25 | 25 | 76
    Mild impairment | 220 | 207 | 205 | 632
    Normal | 126 | 125 | 126 | 377
Chronic Kidney Disease (CKD) Status [Number; unit: participants] — Participant was considered to have CKD if their eGFR was <60 ml/min/1.73 m^2 or urinary albumin:creatinine ratio was >200 mg albumin/g creatinine at Screening.
  participants
    Yes | 25 | 41 | 28 | 94
    No | 347 | 315 | 328 | 990
    Missing | 0 | 1 | 0 | 1
Diabetes Status [Number; unit: participants]
  Yes | 58 | 59 | 71 | 188
  No | 314 | 298 | 285 | 897

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 8 in Trough, Sitting, Clinic Systolic Blood Pressure.
Description: The change in trough systolic blood pressure measured at week 8 or final visit relative to baseline. Systolic blood pressure is the average of the 3 serial trough sitting systolic blood pressure measurements.
Time Frame: Baseline and Week 8.
Population: Full analysis set, all participants that took at least 1 dose of double-blind study drug and have a baseline and post-baseline value, with last observation carried forward.
Measure: Least Squares Mean (Standard Deviation); unit: mmHg
Arm/Group | Azilsartan Medoxomil 20-40mg Plus Chlorthalidone 12.5-25 mg QD | Azilsartan Medoxomil 40-80mg Plus Chlorthalidone 12.5-25 mg QD | Olmesartan Medoxomil 20-40mg/Hydrochlorothiazide 12.5-25mg QD
Number analyzed (Participants) | 363 | 350 | 353
mmHg | -37.6 (0.83) | -38.2 (0.85) | -31.5 (0.84)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 20-40mg Plus Chlorthalidone 12.5-25 mg QD vs Olmesartan Medoxomil 20-40mg/Hydrochlorothiazide 12.5-25mg QD; Analysis of Covariance (ANCOVA) model with treatment as a fixed effect and Baseline as a covariate; Test type: Superiority or Other; p < 0.001, ANCOVA — Statistical significance was set at the 0.05 level per the predefined stepwise testing strategy used; Mean Difference (Final Values) = -6.1, 95% CI 2-sided [-8.4 to -3.8]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 40-80mg Plus Chlorthalidone 12.5-25 mg QD vs Olmesartan Medoxomil 20-40mg/Hydrochlorothiazide 12.5-25mg QD; ANCOVA model with treatment as a fixed effect and Baseline as a covariate; Test type: Superiority or Other; p < 0.001, ANCOVA — Statistical significance was set at the 0.05 level per the predefined stepwise testing strategy used; Mean Difference (Final Values) = -6.7, 95% CI 2-sided [-9.1 to -4.4]

2. Secondary Outcome: Change From Baseline to Week 4 in Trough, Sitting, Clinic Systolic Blood Pressure.
Description: The change in trough systolic blood pressure measured at week 4 relative to baseline. Systolic blood pressure is the average of the 3 serial trough sitting systolic blood pressure measurements.
Time Frame: Baseline and Week 4.
Population: Full analysis set, all participants that took at least 1 dose of double-blind study drug and have a baseline and post-baseline value, with last observation carried forward. Participants who had not achieved target systolic blood pressure/diastolic blood pressure were titrated to the higher dose at week 4.
Measure: Least Squares Mean (Standard Deviation); unit: mmHg
Arm/Group | Azilsartan Medoxomil 20-40mg Plus Chlorthalidone 12.5-25 mg QD | Azilsartan Medoxomil 40-80mg Plus Chlorthalidone 12.5-25 mg QD | Olmesartan Medoxomil 20-40mg/Hydrochlorothiazide 12.5-25mg QD
Number analyzed (Participants) | 360 | 347 | 352
mmHg | -33.0 (0.87) | -34.1 (0.88) | -26.9 (0.88)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 20-40mg Plus Chlorthalidone 12.5-25 mg QD vs Olmesartan Medoxomil 20-40mg/Hydrochlorothiazide 12.5-25mg QD; ANCOVA model with treatment as a fixed effect and Baseline as a covariate; Test type: Superiority or Other; p < 0.001, ANCOVA — Statistical significance was set at the 0.05 level per the predefined stepwise testing strategy used; Mean Difference (Final Values) = -6.1, 95% CI 2-sided [-8.5 to -3.7]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 40-80mg Plus Chlorthalidone 12.5-25 mg QD vs Olmesartan Medoxomil 20-40mg/Hydrochlorothiazide 12.5-25mg QD; ANCOVA model with treatment as a fixed effect and Baseline as a covariate; Test type: Superiority or Other; p < 0.001, ANCOVA — Statistical significance was set at the 0.05 level per the predefined stepwise testing strategy used; Median Difference (Final Values) = -7.2, 95% CI 2-sided [-9.6 to -4.8]

3. Secondary Outcome: Change From Baseline in Trough, Sitting, Clinic Diastolic Blood Pressure
Description: The change in trough diastolic blood pressure measured at week 4 and week 8 relative to baseline. Diastolic blood pressure is the average of the 3 serial trough sitting diastolic blood pressure measurements.
Time Frame: Baseline, Week 4 and Week 8.
Population: Full analysis set , all participants that took at least 1 dose of double-blind study drug and have a baseline and post-baseline value, with last observation carried forward. Participants who had not achieved target systolic blood pressure/diastolic blood pressure were titrated to the higher dose at week 4.
Measure: Least Squares Mean (Standard Deviation); unit: mmHg
Arm/Group | Azilsartan Medoxomil 20-40mg Plus Chlorthalidone 12.5-25 mg QD | Azilsartan Medoxomil 40-80mg Plus Chlorthalidone 12.5-25 mg QD | Olmesartan Medoxomil 20-40mg/Hydrochlorothiazide 12.5-25mg QD
Number analyzed (Participants) | 372 | 357 | 356
mmHg
  Week 4 (n=360; n=347; n=352) | -13.6 (0.49) | -14.2 (0.50) | -10.4 (0.49)
  Week 8 (n=363; n=350; n=353) | -16.1 (0.47) | -16.5 (0.48) | -12.8 (0.48)

4. Secondary Outcome: Change From Baseline in Trough Mean Systolic Blood Pressure Measured by Ambulatory Blood Pressure Monitoring.
Description: The change in trough systolic blood pressure measured at week 4 and week 8 relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. Trough is the average of all measurements recorded from 22 to 24 hours after dosing.
Time Frame: Baseline, Week 4 and Week 8.
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 20-40mg Plus Chlorthalidone 12.5-25 mg QD | Azilsartan Medoxomil 40-80mg Plus Chlorthalidone 12.5-25 mg QD | Olmesartan Medoxomil 20-40mg/Hydrochlorothiazide 12.5-25mg QD
Number analyzed (Participants) | 372 | 357 | 356
mmHg
  Week 4 (n=223; n=227; n=219) | -22.4 (0.95) | -23.6 (0.94) | -17.4 (0.96)
  Week 8 (n=290; n=278; n=281) | -24.9 (0.79) | -26.8 (0.81) | -19.6 (0.80)

5. Secondary Outcome: Change From Baseline in Trough Mean Diastolic Blood Pressure Measured by Ambulatory Blood Pressure Monitoring.
Description: as for outcome 4
Time Frame: Baseline, Week 4 and Week 8.
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 20-40mg Plus Chlorthalidone 12.5-25 mg QD | Azilsartan Medoxomil 40-80mg Plus Chlorthalidone 12.5-25 mg QD | Olmesartan Medoxomil 20-40mg/Hydrochlorothiazide 12.5-25mg QD
Number analyzed (Participants) | 372 | 357 | 356
mmHg
  Week 4 (n=223; n=227; n=219) | -13.4 (0.66) | -14.6 (0.66) | -10.9 (0.67)
  Week 8 (n=290; n=278; n=281) | -14.6 (0.56) | -15.9 (0.57) | -12.0 (0.57)

6. Secondary Outcome: Change From Baseline in 24-hour Mean Systolic Blood Pressure as Measured by Ambulatory Blood Pressure Monitoring.
Description: The change in the 24-hour mean systolic blood pressure at week4 and week 8 relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. The 24-hour mean is the average of all measurements recorded for 24 hours after dosing.
Time Frame: Baseline, Week 4 and Week 8.
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 20-40mg Plus Chlorthalidone 12.5-25 mg QD | Azilsartan Medoxomil 40-80mg Plus Chlorthalidone 12.5-25 mg QD | Olmesartan Medoxomil 20-40mg/Hydrochlorothiazide 12.5-25mg QD
Number analyzed (Participants) | 372 | 357 | 356
mmHg
  Week 4 (n=223; n=227; n=219) | -24.1 (0.81) | -24.4 (0.80) | -18.4 (0.81)
  Week 8 (n=290; n=278; n=281) | -26.4 (0.69) | -27.9 (0.70) | -20.7 (0.70)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 20-40mg Plus Chlorthalidone 12.5-25 mg QD vs Olmesartan Medoxomil 20-40mg/Hydrochlorothiazide 12.5-25mg QD; Statistical analysis for Week 8. ANOVA model with treatment as a fixed effect. Post-baseline p-values are obtained from an ANCOVA model with treatment as a fixed effect and baseline as a covariate; Test type: Superiority or Other; p < 0.001, ANCOVA — Tested at the 0.05 significance level; Mean Difference (Final Values) = -5.6, 95% CI 2-sided [-7.5 to -3.7]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 40-80mg Plus Chlorthalidone 12.5-25 mg QD vs Olmesartan Medoxomil 20-40mg/Hydrochlorothiazide 12.5-25mg QD; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — Tested at the 0.05 significance level; Mean Difference (Final Values) = -7.2, 95% CI 2-sided [-9.1 to -5.2]

7. Secondary Outcome: Change From Baseline in 24-hour Mean Diastolic Blood Pressure Measured by Ambulatory Blood Pressure Monitoring.
Description: The change in the 0 to 24-hours-after-dosing mean diastolic blood pressure measured at Week 4 and Week 8 relative to baseline. . Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. The mean consists of the average of measurements collected over the subsequent 24 hours.
Time Frame: Baseline, Week 4 and Week 8.
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 20-40mg Plus Chlorthalidone 12.5-25 mg QD | Azilsartan Medoxomil 40-80mg Plus Chlorthalidone 12.5-25 mg QD | Olmesartan Medoxomil 20-40mg/Hydrochlorothiazide 12.5-25mg QD
Number analyzed (Participants) | 372 | 357 | 357
mmHg
  Week 4 (n=223; n=227; n=219) | -13.9 (0.51) | -14.4 (0.51) | -10.5 (0.52)
  Week 8 (n=290; n=278; n=281) | -15.1 (0.45) | -16.4 (0.46) | -12.0 (0.46)

8. Secondary Outcome: Change From Baseline in Daytime Mean (6am to 10pm) Systolic Blood Pressure Measured by Ambulatory Blood Pressure Monitoring.
Description: The change in the daytime, while awake (6am to 10pm) mean systolic blood pressure measured at Week 4 and Week 8 relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night Daytime mean is the average of measurements recorded between the hours of 6 AM (inclusive) and 10 PM (exclusive) included in the 24-hour mean calculations.
Time Frame: Baseline, Week 4 and Week 8.
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 20-40mg Plus Chlorthalidone 12.5-25 mg QD | Azilsartan Medoxomil 40-80mg Plus Chlorthalidone 12.5-25 mg QD | Olmesartan Medoxomil 20-40mg/Hydrochlorothiazide 12.5-25mg QD
Number analyzed (Participants) | 372 | 357 | 356
mmHg
  Week 4 (n=223; n=227; n=219) | -24.5 (0.84) | -25.1 (0.83) | -18.9 (0.85)
  Week 8 (n=290; n=278; n=281) | -26.7 (0.72) | -28.4 (0.74) | -21.0 (0.74)

9. Secondary Outcome: Change From Baseline in Daytime Mean (6am to 10pm) Diastolic Blood Pressure Measured by Ambulatory Blood Pressure Monitoring.
Description: The change in the daytime, while awake (6am to 10pm) mean diastolic blood pressure measured at Week 4 and Week 8relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. Daytime mean is the average of measurements recorded between the hours of 6 AM (inclusive) and 10 PM (exclusive) included in the 24-hour mean calculations.
Time Frame: Baseline, Week 4 and Week 8.
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 20-40mg Plus Chlorthalidone 12.5-25 mg QD | Azilsartan Medoxomil 40-80mg Plus Chlorthalidone 12.5-25 mg QD | Olmesartan Medoxomil 20-40mg/Hydrochlorothiazide 12.5-25mg QD
Number analyzed (Participants) | 372 | 357 | 356
mmHg
  Week 4 (n=223; n=227; n=219) | -14.2 (0.53) | -14.7 (0.53) | -10.7 (0.54)
  Week 8 (n=290; n=278; n=281) | -15.3 (0.47) | -16.6 (0.48) | -12.1 (0.48)

10. Secondary Outcome: Change From Baseline in Nighttime Mean (12am to 6am) Systolic Blood Pressure Measured by Ambulatory Blood Pressure Monitoring
Description: The change in the nighttime, while asleep (12am to 6am) mean systolic blood pressure measured at Week 4 and Week 8 to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. Nighttime mean is the average of measurements recorded between the hours of 12 AM (inclusive) and 6 AM (exclusive) included in the 24-hour mean calculations.
Time Frame: Baseline, Week 4 and Week 8.
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 20-40mg Plus Chlorthalidone 12.5-25 mg QD | Azilsartan Medoxomil 40-80mg Plus Chlorthalidone 12.5-25 mg QD | Olmesartan Medoxomil 20-40mg/Hydrochlorothiazide 12.5-25mg QD
Number analyzed (Participants) | 372 | 357 | 356
mmHg
  Week 4 (n=223; n=227; n=219) | -22.3 (0.87) | -21.9 (0.86) | -16.6 (0.88)
  Week 8 (n=290; n=278; n=281) | -25.2 (0.74) | -26.3 (0.75) | -19.7 (0.75)

11. Secondary Outcome: Change From Baseline in Nighttime Mean (12am to 6am) Diastolic Blood Pressure Measured by Ambulatory Blood Pressure Monitoring.
Description: The change in the nighttime, while asleep (12am to 6am) mean diastolic blood pressure measured at Week 4 and Week 8 relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. Nighttime mean is the average (arithmetic mean) of measurements recorded between the hours of 12 AM (inclusive) and 6 AM (exclusive) included in the 24-hour mean calculations.
Time Frame: Baseline, Week 4 and Week 8.
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 20-40mg Plus Chlorthalidone 12.5-25 mg QD | Azilsartan Medoxomil 40-80mg Plus Chlorthalidone 12.5-25 mg QD | Olmesartan Medoxomil 20-40mg/Hydrochlorothiazide 12.5-25mg QD
Number analyzed (Participants) | 372 | 357 | 356
mmHg
  Week 4 (n=223; n=227; n=219) | -13.4 (0.58) | -13.3 (0.58) | -9.6 (0.59)
  Week 8 (n=290; n=278; n=281) | -14.9 (0.51) | -15.8 (0.52) | -11.8 (0.52)

12. Secondary Outcome: Change From Baseline in 12-hr Mean Systolic Blood Pressure Measured by Ambulatory Blood Pressure Monitoring.
Description: The change in the 0 to 12 hours-after-dosing mean Systolic Blood Pressure measured at Week 4 and Week 8 relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night The mean consists of the average (arithmetic mean) of measurements collected at each time frame and includes all observations recorded over the subsequent 12 hours.
Time Frame: Baseline, Week 4 and Week 8.
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 20-40mg Plus Chlorthalidone 12.5-25 mg QD | Azilsartan Medoxomil 40-80mg Plus Chlorthalidone 12.5-25 mg QD | Olmesartan Medoxomil 20-40mg/Hydrochlorothiazide 12.5-25mg QD
Number analyzed (Participants) | 372 | 357 | 356
mmHg
  Week 4 (n=223; n=227; n=219) | -25.0 (0.87) | -25.5 (0.86) | -19.2 (0.88)
  Week 8 (n=290; n=278; n=281) | -27.1 (0.77) | -28.8 (0.78) | -21.1 (0.78)

13. Secondary Outcome: Change From Baseline in 12-hr Mean Diastolic Blood Pressure Measured by Ambulatory Blood Pressure Monitoring.
Description: The change in the 0 to 12 hours-after-dosing mean diastolic blood pressure measured at Week 4 and Week 8 to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. The mean consists of the average (arithmetic mean) of measurements collected at each time frame and includes all observations recorded over the subsequent 12 hours.
Time Frame: Baseline, Week 4 and Week 8.
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 20-40mg Plus Chlorthalidone 12.5-25 mg QD | Azilsartan Medoxomil 40-80mg Plus Chlorthalidone 12.5-25 mg QD | Olmesartan Medoxomil 20-40mg/Hydrochlorothiazide 12.5-25mg QD
Number analyzed (Participants) | 372 | 357 | 356
mmHg
  Week 4 (n=223; n=227; n=219) | -14.4 (0.56) | -14.8 (0.55) | -10.8 (0.56)
  Week 8 (n=290; n=278; n=281) | -15.4 (0.50) | -16.9 (0.51) | -12.1 (0.51)

14. Secondary Outcome: Percentage of Participants Who Achieve a Clinic Systolic Blood Pressure Response, Defined as <140 mm Hg for Participants Without Diabetes or CKD or <130 mm Hg for Participants With Diabetes or CKD
Description: Percentage of participants who achieve a clinic systolic blood pressure response, defined as <140 mm Hg for participants without diabetes or CKD or <130 mm Hg for participants with diabetes or CKD at each time frame relative to baseline.
Time Frame: Baseline, Week 2, Week 4, Week 6 and Week 8.
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Azilsartan Medoxomil 20-40mg Plus Chlorthalidone 12.5-25 mg QD | Azilsartan Medoxomil 40-80mg Plus Chlorthalidone 12.5-25 mg QD | Olmesartan Medoxomil 20-40mg/Hydrochlorothiazide 12.5-25mg QD
Number analyzed (Participants) | 372 | 357 | 356
percentage of participants
  Week 2 (n=343; n=334; n=345) | 60.3 | 57.2 | 44.9
  Week 4 (n=360; n=347; n=352) | 66.1 | 68.9 | 52.3
  Week 6 (n=362; n=350; n=353) | 76.8 | 73.4 | 64.9
  Week 8 (n=363; n=350; n=353) | 76.0 | 76.0 | 64.6

15. Secondary Outcome: Percentage of Participants Who Achieve a Clinic Diastolic Blood Pressure Response, Defined as Defined as <90 mm Hg for Participants Without Diabetes or CKD or <80 mm Hg for Participants With Diabetes or CKD
Description: Percentage of participants who achieve a clinic diastolic blood pressure response, defined as defined as <90 mm Hg for participants without diabetes or CKD or <80 mm Hg for participants with diabetes or CKD at each time frame relative to baseline.
Time Frame: Baseline, Week 2, Week 4, Week 6 and Week 8.
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Azilsartan Medoxomil 20-40mg Plus Chlorthalidone 12.5-25 mg QD | Azilsartan Medoxomil 40-80mg Plus Chlorthalidone 12.5-25 mg QD | Olmesartan Medoxomil 20-40mg/Hydrochlorothiazide 12.5-25mg QD
Number analyzed (Participants) | 372 | 357 | 356
percentage of participants
  Week 2 (n=343; n=334; n=345) | 63.6 | 66.2 | 47.8
  Week 4 (n=360; n=347; n=352) | 71.4 | 73.8 | 58.2
  Week 6 (n=362; n=350; n=353) | 77.9 | 76.9 | 66.9
  Week 8 (n=363; n=350; n=353) | 79.9 | 79.1 | 66.0

16. Secondary Outcome: Percentage of Participants Who Achieve a Clinic Diastolic AND Systolic Blood Pressure Response, Defined as <140/90 mm Hg for Participants Without Diabetes or Chronic Kidney Disease (CKD) or <130/80 mm Hg for Participants With Diabetes or CKD
Description: Percentage of participants who achieve both a clinic diastolic blood pressure response, defined as <140/90 mm Hg for participants without diabetes or chronic kidney disease (CKD) or <130/80 mm Hg for participants with diabetes or CKD at each time frame relative to baseline.
Time Frame: Baseline, Week 2, Week 4, Week 6 and Week 8.
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Azilsartan Medoxomil 20-40mg Plus Chlorthalidone 12.5-25 mg QD | Azilsartan Medoxomil 40-80mg Plus Chlorthalidone 12.5-25 mg QD | Olmesartan Medoxomil 20-40mg/Hydrochlorothiazide 12.5-25mg QD
Number analyzed (Participants) | 372 | 357 | 356
percentage of participants
  Week 2 (n=343; n=334; n=345) | 51.3 | 48.5 | 35.9
  Week 4 (n=360; n=347; n=352) | 58.1 | 61.4 | 44.6
  Week 6 (n=362; n=350; n=353) | 68.8 | 65.4 | 55.5
  Week 8 (n=363; n=350; n=353) | 69.4 | 68.9 | 54.7

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are adverse events that started on or after the first dose of double-blind study drug and no more than 14 days (or 30 days for a serious adverse event) after the last dose of double-blind study drug.
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Azilsartan Medoxomil 20-40mg Plus Chlorthalidone 12.5-25 mg QD | Azilsartan Medoxomil 40-80mg Plus Chlorthalidone 12.5-25 mg QD | Olmesartan Medoxomil 20-40mg/Hydrochlorothiazide 12.5-25mg QD
Serious Adverse Events (participants affected / at risk) | 4/372 | 8/357 | 6/356
Other Adverse Events (participants affected / at risk) | 66/372 | 72/357 | 56/356
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Azilsartan Medoxomil 20-40mg Plus Chlorthalidone 12.5-25 mg QD (N=372) | Azilsartan Medoxomil 40-80mg Plus Chlorthalidone 12.5-25 mg QD (N=357) | Olmesartan Medoxomil 20-40mg/Hydrochlorothiazide 12.5-25mg QD (N=356)
Cardiac arrest (Cardiac disorders) | 0 | 1 | 1
Coronary artery disease (Cardiac disorders) | 0 | 0 | 1
Diastolic dysfunction (Cardiac disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0
Epigastric discomfort (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 1
Generalised oedema (General disorders) | 0 | 1 | 0
Systemic inflammatory response syndrome (General disorders) | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1 | 1
Gastroenteritis (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0
Viral infection (Infections and infestations) | 0 | 1 | 0
Heat exhaustion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 0
Troponin increased (Investigations) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1
Shock (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Azilsartan Medoxomil 20-40mg Plus Chlorthalidone 12.5-25 mg QD (N=372) | Azilsartan Medoxomil 40-80mg Plus Chlorthalidone 12.5-25 mg QD (N=357) | Olmesartan Medoxomil 20-40mg/Hydrochlorothiazide 12.5-25mg QD (N=356)
Blood creatinine increased (Investigations) | 36 | 44 | 25
Dizziness (Nervous system disorders) | 25 | 24 | 20
Headache (Nervous system disorders) | 14 | 14 | 18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No publication related to study results will be published prior to publication of a multi-center report submitted for publication within 18 months after conclusion or termination of a study at all study sites. Results publications will be submitted to sponsor for review 60 days in advance of publication. Sponsor can require removal of confidential information unrelated to study results. Sponsor can embargo a proposed publication for another 60 days to preserve intellectual property.